CLINICAL TRIAL: NCT02218866
Title: The Effect of Bariatric Surgery on Peripheral Nerve Function and Axonal Regeneration
Acronym: BAR
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Gordon Smith, Professor, University of Utah
Other Study IDs: BAR-UofU
Record Dates: First submitted 2014-08-04; First posted 2014-08-18 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2016-08

CONDITIONS: Peripheral Neuropathy; Obesity
Keywords: Bariatric surgery; Obesity; Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: All participants will be examined by a neurologist to test sensation, reflexes, and strength and complete a few questionnaires. Tests will be performed to measure nerve function and small punch skin biopsies will be taken to assess nerve fiber density. Blood and urine tests will measure various markers of interest. Participants will be seen before and after their bariatric surgery.
- Group 2: In addition to the procedures described for Group 1, participants in Group 2 will have the following procedures:
  * During bariatric surgery, a small biopsy from the liver and abdominal fat will be taken to examine how fat is processed within the body.
  * At the first visit, after a skin biopsy is taken, a small capsaicin patch will be placed on the lower thigh. The patch will remain in place for 48 hours and will cause the nerves in the immediate area to pull back from the skin. A biopsy will be taken from the patch area 48 hours, 1 month, and 3 months after the initial biopsy. This procedure will be repeated after surgery.
  * MRIs may be performed before and after bariatic surgery.
  * Participants may be asked to complete additional tests to evaluate nerve function
- Group 3: Group 3 will comprise of individuals who are not overweight. Participants in this group will undergo a similar evaluation to Group 2.

SUMMARY:
The goal of this research is understand if obesity is a major factor for neuropathy development in patients with and without Type 2 diabetes. This study will examine the relationship between weight, metabolism, and nerve function and regeneration.

DETAILED DESCRIPTION:
Peripheral neuropathy causes progressive injury to the longest nerves of the body, starting in the toes, then progressing slowly up the leg. Neuropathy often causes pain, numbness, and weakness if the feet and can lead to reduced mobility, foot ulcers, and even amputation. The most common cause is diabetes, but work at the University of Utah finds that prediabetes and other consequences of obesity, including abnormal cholesterol levels, may be associated with neuropathy. Research has shown that these risk factors may damage nerves and interfere with the ability of nerves to grow back after an injury.

This study aims to

1. characterize peripheral nerve function and cutaneous nerve structure in obese bariatric surgery candidates;
2. evaluate peripheral nerve regeneration capacity (and other nerve function measures) before and after bariatric surgery in obese subjects with no or mild neuropathy;
3. examine the relationship between ectopic lipid accumulation, lipotoxic mediators, neuropathy and regeneration capacity in surgical candidates before and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Subjects must fulfill criteria for bariatric surgery.

Exclusion Criteria:

* History of foot ulceration or neurogenic arthropathy
* Family history of non-diabetic neuropathy in a first-degree family member.
* Presence of any disease known to be associated with peripheral neuropathy including but not limited to vitamin deficiency, toxin exposure, paraproteinemia, heavy alcohol use, hepatitis C, HIV.
* Coumadin use.
* Inability to understand or cooperate with the procedures of the trial.
* Known history of sensitivity to capsaicin products.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through bariatric surgery clinics in the local area.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2012-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in reinnervation capacity | 4 - 1 months prior to bariatric surgery, compared to 9 - 12 months after surgery

SECONDARY OUTCOMES:
Change in Utah Early Neuropathy Scale (UENS) | Baseline to 12 months after bariatric surgery
Change in Nerve Conduction Study measures | Baseline to 12 months after bariatric surgery
  Nerve Conduction Study is a procedure routinely used in the diagnosis of neuropathy. Measures will include Sural sensory and Peroneal motor amplitudes and conduction velocities.
Change in nerve fiber density | Baseline to 12 months after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: A. Gordon Smith, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States